CLINICAL TRIAL: NCT02725489
Title: Pilot Study of Durvalumab (MEDI4736) in Combination With Vigil in Advanced Women's Cancers
Brief Title: Pilot Study of Durvalumab and Vigil in Advanced Women's Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mary Crowley Medical Research Center (Other)
Collaborators: Gradalis, Inc. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-06; CL-PTL 124 (Other: Gradalis); ESR-15-11306 (Other: Astra Zeneca)
Record Dates: First submitted 2016-03-23; First posted 2016-04-01 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Uterine Cancer; Cervical Cancer; Endometrial Cancer
Keywords: Vigil; durvalumab; MEDI4736; PD-L1; anti PD-L1; immunotherapy; PD-L1 inhibitor; breast cancer; ovarian cancer; fallopian tube cancer; primary peritoneal cancer; uterine cancer; cervical cancer; endometrial cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — FANG vaccine; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Cohort 1: 1x10^6 cells Vigil (Experimental): The first part will be a safety run-in comprised of 2 cohorts that will use a 3 + 3 design to determine the Vigil dose in Part 2. Cohort 1 will receive a low dose of Vigil (1x10^6 cells/intradermal (ID) injection) in combination with durvalumab (1500 mg (if > 30 kg) IV over 60 minutes) every 4 weeks.
  Interventions: Biological: Vigil; Drug: Durvalumab
- Part 1 Cohort 2: 1x10^7 cells Vigil (Experimental): Cohort 2 will receive Vigil at 1x10^7 cells/ID injection and durvalumab (1500mg (if > 30 kg) IV over 60 minutes) every 4 weeks.
  Interventions: Biological: Vigil; Drug: Durvalumab
- Part 1 Cohort -1: 1x10^5 cells Vigil (Experimental): If needed, Cohort -1 will be used which will receive Vigil at 1x10^5 cells/ID injection and Durvalumab (1500mg (if > 30 kg) IV over 60 minutes) every 4 weeks.
  Interventions: Biological: Vigil; Drug: Durvalumab

INTERVENTIONS:
Biological: Vigil — Vigil is made up of irradiated autologous tumor cells which have been electroporated ex vivo with the Vigil plasmid designed to suppress expression of both the TGFβ1 and TGFβ2 proteins while simultaneously expressing rhGMCSF protein.
  Other Names: bi-shRNAfurin and GMCSF Autologous Tumor Cell Immunotherapy; FANG
Drug: Durvalumab — A human immunoglobulin G1 kappa (IgG1κ) monoclonal antibody directed against programmed cell death ligand 1 (PD-L1)
  Other Names: MEDI4736

SUMMARY:
In this study, the researchers want to learn more about Vigil and durvalumab in advanced women's cancers: 1) how much of Vigil in combination with durvalumab (MEDI4736) can be given with an acceptable level of side effects, 2) the effects of Vigil and durvalumab in combination (good and bad), 3) if Vigil will cause changes in cancer cells that may help durvalumab attack the cancer, and 4) whether or not Vigil and durvalumab will slow your cancer or stop your cancer from getting worse.

Combining Vigil with durvalumab will allow the former to induce (or increase) the infiltration of activated T cells into tumors, and in addition, to enhance PD-L1 (programmed cell death ligand 1) expression. Consequently, the response rate of historically low or un-responsive cancer will be increased with the combination of Vigil and anti PD-L1.

DETAILED DESCRIPTION:
This is an open label pilot study to evaluate the safety, tolerability, and efficacy of the combination of Vigil autologous tumor cell immunotherapy and durvalumab PD-L1 inhibitor in patients with locally advanced or metastatic women's cancers, inclusive, but not limited to breast, ovarian, cervical, uterine, fallopian, primary peritoneal, and endometrial regardless of the number of prior therapies.

This will be a 2-part study. The first part will be a safety run-in comprised of 2 cohorts that will use a 3 + 3 design to determine the Vigil dose in Part 2. Patients in Cohort 1 will receive a low dose of Vigil (1x10^6 cells/intradermal (ID) injection) in combination with durvalumab (1500 mg (if > 30 kg) IV over 60 minutes) every 4 weeks. Patients in Cohort 2 will receive Vigil at 1x10^7 cells/ID injection and durvalumab (1500mg (if > 30 kg) IV over 60 minutes) every 4 weeks. If needed, patients in Cohort -1 will receive Vigil at 1x10^5 cells/ID injection and durvalumab (1500mg (if > 30 kg) IV over 60 minutes) every 4 weeks. The enrollment of the first two patients in each Cohort of Part 1 will be staggered by 2 weeks. In Part 2 of the study, patients meeting study eligibility criteria will receive Vigil at the dose determined in Part 1 and durvalumab (1500mg (if > 30 kg) IV over 60 minutes) every 4 weeks. As of March 13, 2018, Part 2 of the study will not be initiated due to limited enrollment. Currently only patients who have Vigil immunotherapy available from Gradalis protocol CL-PTL-119 may be considered for the study.

Radiological assessment of tumor response or alternative assessments of disease status should be performed at screening, Cycle 3 and every 2 cycle thereafter, and end of treatment (EOT) using RECIST 1.1 and investigator assessment as applicable. Tumor biopsy for correlative studies including but not limited to scoring of tumor infiltrating lymphocyte (TIL) and PD-1 / PD-L1 expression analysis should be obtained at tissue procurement and at Cycle 3, and optional biopsies thereafter if the patient has accessible tissue. Peripheral blood mononuclear cells (PBMC) for correlative studies should be obtained at pre-procurement if applicable, and prior to study regimen administration at Cycle 1, Cycle 3, Cycle 5 and EOT. Patient survival will be followed for 1 year after last dose of either Vigil or durvalumab.

ELIGIBILITY:
Inclusion Criteria:

Tissue Procurement Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document for tissue harvest
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Histologically or cytologically confirmed diagnosis of women's cancer, inclusive, but not limited to breast, ovarian, fallopian tube, primary peritoneal, uterine, cervical, endometrial, that is locally advanced or metastatic for which the projected response rate to durvalumab is 15% or less.
* Female patients age ≥ 18 years
* No prior Vigil immunotherapy
* Treatment-naïve or refractory (no response to checkpoints) / resistant (initial response but relapse) to PD-1 or PD-L1 inhibitor therapy
* ECOG Performance Status ≤ 1
* Estimated survival ≥ 6 months
* Planned standard of care surgical procedure (e.g., tumor biopsy or palliative resection or thoracentesis) and expected availability of a cumulative mass of ~10-30 grams tissue ("golf-ball" size) or pleural fluid estimated volume ≥ 500mL (must be primary tap) for immunotherapy manufacture.
* One lesion not previously irradiated nor intended for vaccine manufacture, which can be biopsied with minimal invasion and measurable at baseline as per RECIST 1.1 guidelines (performed prior to biopsy) or 2 lesions not previously irradiated nor intended for vaccine manufacture, one of which can be biopsied with minimal invasion and the other of which is measurable at baseline as per RECIST 1.1 guidelines. If the only such target lesion has previously been irradiated it must have shown unequivocal evidence of disease progression following completion of radiation therapy. Alternative methods of disease assessment, e.g. measurement of tumor markers or ascites/pleural fluid, may be considered by the Sponsor on a case-by-case basis.
* Provision of tumor tissue sample (archived or fresh) to allow for PD-L1 expression analysis

Study Enrollment Inclusion Criteria:

* Successful manufacturing of at least 4 vials of Vigil.
* Ability to understand and the willingness to sign a written informed consent document
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Estimated survival of ≥ 6 months
* Provision of tumor tissue sample (archived or fresh) in a quantity sufficient to allow for PD-L1 expression analysis (if not already obtained during tissue procurement under this protocol), and after entry, a portion of Vigil harvested tissue
* If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, complete hysterectomy, or surgery for gynecological cancer) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
* Adequate organ and bone marrow function as defined below:

  1. Absolute neutrophil count (ANC) > 1.5 × 10^9/L (1500 per mm^3)
  2. Platelets > 100 × 10^9/L (100,000 per mm^3)
  3. Hemoglobin ≥ 9.0 g/dL (5.59 mmol/L)
  4. Creatinine clearance (CrCL) > 50 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance:

     Females: CrCL (mL/min) = Weight (kg) × (140 - Age) × 0.85 / 72 × serum creatinine (mg/dL)
  5. Serum bilirubin ≤ 1.5 × upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of evidence of hemolysis or hepatic pathology) who will be allowed in consultation with their physician.
  6. AST and ALT ≤ 2.5 × ULN in patients with no liver metastasis
  7. AST or ALT ≤ 5 × ULN in patients with liver metastasis
  8. TSH within institutional limits. If TSH is greater or less than institutional limits patients may participate if their T4 is within normal limits (WNL); patients may be on a stable dose of replacement thyroid medication; dose adjustments are allowed if needed.
* Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery

  1. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade > 2 or better
  2. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the IPs may be included (e.g., hearing loss) after consultation with the Medical Monitor
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) prior to tissue procurement and at least 21 days prior to the first dose of study drug (at least 21 days prior to the first dose of study drug for subjects who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 week for nitrosourea or mitomycin C). (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required.)

Exclusion Criteria:

Tissue Procurement Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational (noninterventional) clinical study or the follow-up period of an interventional study.
* Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily for < 30 days duration.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent.
* Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 5 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
* History of brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 4 months.
* Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids (unless within the protocol allowed doses).
* Known history of allergies or sensitivities to gentamicin, Durvalumab, or any excipient.
* History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Known HIV or acute or chronic Hepatitis B or C infection.
* History of pneumonitis or interstitial lung disease.
* History of organ transplant that requires therapeutic immunosuppression
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of Peptic Ulcer Disease or gastritis
* History of primary immunodeficiency
* History of leptomeningeal carcinomatosis
* Known history of previous clinical diagnosis of tuberculosis
* Previous allogeneic bone marrow transplant
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment in the present study

Study Enrollment Exclusion Criteria:

* Palliative radiotherapy within 3 weeks of start of study therapy. Limited field of radiation for palliation greater than 3 weeks prior to the first dose of study treatment is allowed:

  1. Provided the lung is not in the radiation field
  2. Provided irradiated lesion(s) cannot be used as target lesions
* Receipt of steroid therapy during the last 2 weeks prior to study enrollment and study treatment start.
* Post-surgery complication that in the opinion of the treating investigator would interfere with the patient's study participation or not be in the best interest of the patient to participate
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of Vigil or Durvalumab. NOTE: Subjects, if enrolled, should not receive live vaccine during the study and 30 days after the last dose of both drugs.
* Post-surgery complication that in the opinion of the treating investigator would interfere with the patient's study participation or make it not in the best interest of the patient to participate
* Participation in another clinical study with an investigational product during the last 3 weeks
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
* Female subjects who are pregnant, breast-feeding or of reproductive potential who are not employing an effective method of birth control defined in the protocol (section 7.6)
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent AEs of Vigil + Durvalumab | Up to 90 days after last dose of study treatment
  The safety evaluation will include collection of AEs, SAEs and changes from baseline in laboratory evaluations, vital signs, ECGs and physical exams. AEs will be graded according to the NCI CTCAE v4.03.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 12 months after start of study treatment
  The ORR will be estimated in patients with measurable disease, along with its exact binomial 95% confidence interval.
Disease status | Up to 12 months after start of study treatment
  Disease status will be summarized based on tumor markers or ascites/pleural fluid in patients with non-measurable disease
IFNγ-ELISPOT conversion rate (negative to positive) during on-study treatment | 12 weeks after start of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Mary Crowley Cancer Research
Locations (1):
- Mary Crowley Cancer Research Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No